CLINICAL TRIAL: NCT05822466
Title: A Remotely Delivered Tai Ji Quan Intervention to Reduce Incidence of Falls in High Risk Community-Dwelling Older Adults
Brief Title: Virtual Tai ji Quan Exercise to Prevent Falls in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AG081206 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Accidental Fall

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual tai ji quan (Active Comparator): Participants participating are intervened with practice and drills of tai ji quan forms and associated movements. Training focuses on lower-extremity strength, postural control, and mobility, with an emphasis on weight bearing and weight shifting, extending and controlling the body's center of mass over its base of support; self-induced movement perturbation; gait preparation, initiation, locomotion, and termination; and sensory integration. The exercise training also emphasizes connecting tai ji quan forms to transitional movements that are associated with performing daily activities. Each session includes brief movement-based warm-ups and light breathing cool-down exercises.
  Interventions: Behavioral: Virtual tai ji quan: moving for better balance intervention (V-TJQMBB)
- Virtual multimodal exercise (Active Comparator): Participants participating are intervened with a multicomponent exercise program that involves light walking, strength, postural control, and flexibility exercises. Walking exercises include amble forward and backward walk, long strides, heel-toe walking, narrow- and wide-base walking, and sidestepping. Strength training includes single- and multi-joint exercises such as semi-squats, lunging forward and sideways, and toe stands that involve exercising ankle dorsiflexors, knee extensors, and hip abductors. Balance training involves semi-tandem foot-standing, heel-toe and line walking, single-leg standing, alternation of the base of support, weight transfers, toe and heel movements, and various reaching and stretching movements away from the center of the base of support. Flexibility exercises include a static stretching routine of major upper and lower body muscle groups. Each session includes brief movement-based warm-ups and light breathing cool-down exercises.
  Interventions: Behavioral: Virtual multimodal exercise intervention (V-Multimodal)

INTERVENTIONS:
Behavioral: Virtual tai ji quan: moving for better balance intervention (V-TJQMBB) — This intervention involves a tai ji quan exercise program, named tai ji quan: moving for better balance
  Other Names: V-TJQMBB
  Arms: Virtual tai ji quan
Behavioral: Virtual multimodal exercise intervention (V-Multimodal) — This intervention involves a multimodal exercise program that consists of balance, strength, light walking, and stretching exercises
  Other Names: V-Multimodal
  Arms: Virtual multimodal exercise

SUMMARY:
To examine two different exercise programs in reducing incidence of falls among community-dwelling older adults

DETAILED DESCRIPTION:
This is a randomized controlled trial aimed at determining the effectiveness of a virtual and home-based tai ji quan intervention vs. a virtual and home-based multimodal exercise intervention in reducing incidence of falls among community-dwelling older adults at high risk of falling

ELIGIBILITY:
Inclusion Criteria:

* age between 65 and 90 years and
* having had 1 or more falls in the preceding 12 months or having a score ≥12 seconds on the Timed Up&Go (TUG) test.

Exclusion Criteria:

* showing a diagnosis of dementia or significant cognitive impairment, as indicated by a score of <24 on the Mini Mental State Evaluation (MMSE, range: 0-30);
* being unable to ambulate independently for household distances; (c) having no medical clearance;
* having participated in any regular and structured tai ji quan-based or multicomponent exercise programs (≥2 times weekly) in the preceding 6 months;
* having any physical condition that would preclude participation in moderate-intensity exercise; and
* being unwilling to commit to the duration of the intervention or accept group assignment.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported number of falls | Monthly, baseline to 6 months
  This measure will reflect change in the incidence of falls as a result of intervention. Study participants will be given a falls calendar to record number of falls at home. Falls are defined as "when you land on the floor or the ground, or fall and hit objects like stairs or pieces of furniture, by accident." This information will be ascertained monthly via a phone call by study assessors

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, 4 months, 6 months, and 12 months
  This measure reflects change in lower extremity function with intervention. This is measured by SPPB which involves three functional tasks: static balance, gait speed, and getting in and out of a chair, with scores ranging from 0 (worst performance) to 12 (best performance).
Timed up and Go (TUG) | Baseline, 4 months, 6 months, and 12 months
  Reflects change in mobility performance with intervention. This is measured by TUG (measured in seconds) which assesses mobility and fall risk. The test measures the time taken by an individual to stand up from a standard chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down. Lower scores represent better lower extremity physical function.
30-second chair stand | Baseline, 4 months, 6 months, and 12 months
  Reflects change in lower-extremity strength with intervention. This is measured by a 30-second chair stand test.
Dual-task walking | Baseline, 4 months, 6 months, and 12 months
  Reflects change in dual-task costs in gait speed with intervention. The TUG test protocol will be repeated under a dual-task condition where the participant is asked to walk while performing an arithmetic task. Lower scores on this walk indicate better performance. Dual-task walking cost is defined as the difference between single- and dual-task walking speed, expressed in percentage, with less negative values representing improvement in dual-task walking speed relative to single-task walking.
Montreal Cognitive Assessment (MoCA) | Baseline, 4 months, 6 months, and 12 months
  Reflects change in global cognitive function. This is measured by MoCA which measures cognitive function of multiple domains (attention/concentration, executive functions, short term memory, language, visuospatial abilities, orientation to time and place). MoCA has a total score that ranges from 0 to 30, with higher scores representing better cognitive functioning.
Trail Making (A, B) | Baseline, 4 months, 6 months, and 12 months
  Reflects change in executive function with intervention. This is measured by Trail Making Test (TMT) which consists of two parts (A and B). In Part A, the participant is asked to count the number (1 through 25) off the screen out loud as quickly as possible. In Part B, the participant is asked to recite numbers and letters in an alternating sequence (1-A-2-B-3-C . . . 12-L) as quickly as possible. Errors are corrected immediate with the clock running. For Parts A and B, scoring is expressed in terms of the time (in seconds) to completion. The difference in time taken to complete Part B versus Part A is calculated to form a measure of executive function, with smaller difference scores indicating better executive function.
Category Fluency | Baseline, 4 months, 6 months, and 12 months
  Reflects change in memory with intervention. This is measured by a category fluency test in which the participant is asked to generate the names of as many animals as possible in 60 seconds.
Forward Digit Span | Baseline, 4 months, 6 months, and 12 months
  Reflects change in attention with intervention. This is measured by Forward Digit Span test. During the test, the participant is asked to repeat a series of digits in the order given. The maximum raw score is 16, with higher scores indicating better attention.
Backward Digit Span | Baseline, 4 months, 6 months, and 12 months
  Reflects change in short-term working memory with intervention. This is measured by Backward Digit Span test. During the test, the participant is asked to repeat a series of digits in reverse order. The maximum raw score is 16, with higher scores indicating better memory.
Proportion of fallers | At 6 months
  Number of fallers from the participants in each intervention group

OTHER OUTCOMES:
Activity-specific Balance Confidence (ABC) | Baseline, 4 months, 6 months, and 12 months
  Reflects change in the perceptions of balance with intervention. This is measured by the ABC scale which assesses one's confidence in performing various activities of daily living without compromising one's balance. It includes such items as picking up an object from the floor, standing on a chair to reach, and walking on icy sidewalks. The scale contains 16 items scored on a range from 0% to 100% (0 indicating no confidence and 100 indicating full confidence).
Pittsburgh Sleep Quality Index | Baseline, 4 months, 6 months, and 12 months
  Reflects change in quality of sleep with intervention. This is measured by the Pittsburgh Sleep Quality Index which includes seven indices: subjective quality, latency (i.e., time needed to fall asleep), duration (i.e., number of hours of actual sleep per night), efficiency (i.e., total sleep time divided by time in bed, converted to a score of 0-3), sleep disturbances (e.g., waking up in the middle of the night and the like), use of sleep medication, and daytime dysfunction (e.g., having difficulty staying awake during the day). Each of the component scores ranges from 0 to 3, with the PSQI global score ranging from 0 to 21 points, with higher scores indicating poorer sleep quality.
Geriatric Depression Scale | Baseline, 4 months, 6 months, and 12 months
  Reflects change in the level of depression with intervention. This is measured by GDS. The 15-item version of the GDS will be used with the scores ranging from 0 to 15. A score of 0 to 4 is considered to be within the normal range, 5 to 9 indicates mild depression, and a score of 10 or more indicates moderate to severe depression.
EuroQol EQ-5D | Baseline, 4 months, 6 months, and 12 months
  Reflects change in quality of life with intervention. This is measured by EuroQol EQ-5D which assesses health status in five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is measured at three levels: no problems (coded as 1), some problems (2), and extreme problems (3). An EQ-5D utility score will be calculated for each participant based on the U.S. population-based (preference-weighted) health index scores on a scale ranging from less than 0 (worst health state) to 1.0 (best or perfect health state).
Frailty Questionnaire | Baseline, 4 months, 6 months, and 12 months
  Reflects change in frailty with intervention. Frailty is measured by the Frailty Questionnaire which assesses 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of Weight. The scale scores range from 0 to 5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status
International Physical Activity Questionnaire | Baseline, 4 months, 6 months, and 12 months
  Reflects change in physical activity with intervention. Total weekly minutes spent in vigorous physical activity (PA) and moderate PA will be measured. Two self-report PA measures will be calculated: total weekly minutes of vigorous + moderate PA in bouts of ≥10 min, excluding walking (MVPA) and total weekly minutes of walking in bouts of ≥10 min (Walk). We will report Total PA (MVPA + Walk), which is conceptually the same construct as accelerometry MVPA in ≥10 min bouts.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Institute, Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes